CLINICAL TRIAL: NCT02383264
Title: Splanchnic Oxygenation Patterns in Response to the First Enteral Feed in Preterm Infants: Prediction of Feeding Tolerance and Correlation With Abnormal Antenatal Doppler.
Brief Title: Splanchnic Oxygenation After the First Enteral Feed in Preterm Infants: Prediction of Feeding Tolerance.
Acronym: NIRS-SO
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Luigi Corvaglia, Associate Professor, University of Bologna (Italy), IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: SO-2015-NIRS; 122/2012/U/Oss (Other: Ethic Committee of St. Orsola-Malpighi University Hospital)
Record Dates: First submitted 2015-03-04; First posted 2015-03-09 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Necrotizing Enterocolitis; Very Low Birth Weight Infants
Keywords: feeding intolerance; preterm infants; near infrared spectroscopy
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- feeding intolerance: Development of feeding intolerance, defined as enteral feeding withholding for at least 1 day due to the onset ofgastrointestinal clinical symptoms
- normal feeding tolerance: no evidence of feeding intolerance during the hospitalization

SUMMARY:
Enteral nutrition of preterm and intrauterine growth-restricted (IUGR) infants is still a challenge for neonatologists. Due to the immaturity of the gastrointestinal tract, preterm infants are at high risk of developing feeding intolerance (FI) or necrotizing enterocolitis (NEC), which is the most feared gastrointestinal complication of prematurity. The occurrence of FI often prompts clinicians to withhold, decrease or discontinue enteral feeds; thus, the establishment of an adequate early enteral nutrition is frequently hampered. Early identification of preterm infants at high risk for gastrointestinal complications could help clinical decisions on the introduction and the advancement of enteral feeding.

Near-infrared spectroscopy (NIRS) provides a non-invasive monitoring of regional oxygen saturation (rSO2). A significant correlation between lower abdominal rSO2 values in the first week of life and subsequent NEC development has been reported. To date, however, splanchnic oxygenation patterns in response to the first bolus feed and possible correlations with subsequent FI development have not been yet established.

This observational prospective study aims:

* to assess abdominal rSO2 patterns in response to the first bolus feed;
* to evaluate possible correlations with subsequent development of gastrointestinal complications.

DETAILED DESCRIPTION:
Enteral nutrition of preterm and intrauterine growth-restricted (IUGR) infants remains a major challenge for neonatologists. Early introduction of minimal enteral feeding (MEF) enhances gut hormones release, reduces the intestinal permeability and improves the motility of the intestinal tract, thus promoting gut functional maturation. Due to gastrointestinal immaturity, however, preterm infants are likely to develop clinical symptoms of feeding intolerance (FI), such as abdominal distention, vomiting, abundant and/or bilious gastric residuals, occult or gross bloody stools. FI could represent an early sign of necrotizing enterocolitis (NEC), the most feared gastrointestinal complication of prematurity. The occurrence of FI often prompts neonatologists to withhold, decrease or discontinue enteral feeds, thus hampering the establishment of an adequate early enteral nutrition.

Early identification of preterm infants at high risk of gastrointestinal complications could help clinical decisions on the introduction and the advancement of enteral feeding. The administration of the first feed in healthy preterm infants leads to a post-prandial increase of superior mesenteric artery (SMA) blood flow, detected by Doppler ultrasound. A significant correlation between early feeding tolerance and increased SMA blood flow velocity has been further observed one hour after the first feed.

Near-infrared spectroscopy (NIRS) provides a non-invasive monitoring of regional oxygen saturation (rSO2) and has been previously used to evaluate mesenteric perfusion in preterm infants at increased risk for intestinal complications. Abdominal rSO2 detected by NIRS has been shown to effectively reflect mesenteric blood flow changes. A significant correlation between lower abdominal rSO2 values in the first week of life and subsequent NEC development has been recently observed in a cohort of preterm infants, confirming previous data from animal models.

Current evidences on the role of NIRS monitoring in predicting FI development are still limited. To date, indeed, splanchnic oxygenation patterns in response to the first bolus feed and possible correlations with subsequent FI development have not been established yet.

The aim of this study is to assess abdominal rSO2 patterns in response to the first bolus feed and to evaluate possible correlations with the development of gastrointestinal complications.

Infants admitted to the Neonatal Intensive Care Unit (NICU) are consecutively enrolled in the study if fulfilling the following criteria: gestational age ≤34 weeks, stable clinical conditions, availability of antenatal Doppler data.

Exclusion criteria are:

* Enteral feeding prior to the enrollment
* Major congenital abnormalities
* Central nervous system diseases
* Hypoxic injury
* Hemodynamic instability, hypotension, patent ductus arterioles, anemia, sepsis or other infections at time of the first feed.
* Antenatal Doppler impairment.

Written, informed consent to participate in the study is obtained from the parents/legal guardians of each infant before enrollment.

During the first feed administration, the enrolled infants undergo a continuous monitoring of cerebral and splanchnic rSO2 by means of an INVOS 5100 oximeter. NIRS recording is performed from 30 minutes before to 3 hours after feeding administration. Cerebral and splanchnic rSO2 are recorded every 5 seconds. Baseline values are defined by the mean of the 15 minutes before the meal; values recorded after feeding administration are clustered into 5-minute intervals.

Feeding intolerance is defined as enteral feeding withholding for at least 1 day due to the onset of gastrointestinal symptoms.

Patients' characteristics (including gestational age, birth weight, tolerance to enteral feeds during hospitalization) are recorded in a specific case report form at the time of enteral feeding introduction and before discharge.

In relation to their clinical characteristics, the enrolled infants are retrospectively allocated into 2 groups:

* Group 1: infants developing FI during the hospitalization;
* Group 2: infants not developing FI during the hospitalization;

Data are analyzed using IBM SPSS Statistic version 20.0.0 (IBM Corporation, IBM Corporation Armonk, New York, United States). Clinical characteristics in the study groups are compared by t-test for continuous variables and chi-square test for categorical variables. Mann-Whitney U test is used to compare abdominal rSO2 patterns in response to the first feed between groups 1 and 2. A multivariate analysis is also performed to assess the effect of possible confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≤34 weeks
* Stable clinical conditions

Exclusion Criteria:

* Any enteral feeding prior to the enrollment.
* Major congenital abnormalities
* Central nervous system diseases
* Hypoxic injury
* Hemodynamic instability, hypotension, patent ductus arterioles, anemia, sepsis or other infections at time of first feed.
* Antenatal Doppler impairment.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Due to the exploratory nature of this study, at least 60 preterm infants admitted to the Neonatal Intensive Care Unit of Sant'Orsola-Malpighi University Hospital and fulfilling the inclusion criteria are going to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Increase/reduction of abdominal rSO2 values after the first enteral feed in infants at high risk of feeding intolerance. | 3.5 hours
  Increase/reduction of abdominal rSO2 values in response to the first enteral feed in infants who have further developed feeding intolerance during their hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi T Corvaglia, Prof, Principal Investigator — S. Orsola-Malpighi Hospital, University of Bologna
Locations (1):
- Neonatal Intensive Care Unit of the S.Orsola-Malpighi Hospital, Bologna, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Corvaglia L, Martini S, Battistini B, Rucci P, Faldella G, Aceti A. Splanchnic Oxygenation at First Enteral Feeding in Preterm Infants: Correlation With Feeding Intolerance. J Pediatr Gastroenterol Nutr. 2017 Apr;64(4):550-554. doi: 10.1097/MPG.0000000000001308. PMID 27467111